CLINICAL TRIAL: NCT06968299
Title: Effect of ExoBDNF Lactic Acid Bacteria Supplement on Cognitive Functions, Sleep and Psychological Outcomes: An Open-label Trial
Brief Title: Effect of ExoBDNF Lactic Acid Bacteria Supplement on Cognitive Functions, Sleep and Psychological
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-ExoBDNF-1
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Functions Perceptual Disturbances; Cognitive Function Abnormal; Sleep; Psychological
Keywords: Probiotics; ExoBDNF; Cognitive functions
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExoBDNF SWP-CGPA01 (Pediococcus acidilactici)Capsules (Experimental): ExoBDNF is the product name of SWP-CGPA01 Pediococcus acidilactici, which is listed as a food-usable strain in Taiwan, China, Europe and the United States. The strain has been deposited in the National Collection of Industrial Food and Marine Bacteria (NCIMB) in the United Kingdom, and the strain number is NCIMB 44102. 1.0 x 1010 CFU SWP-CGPA01 freeze-dried powder (production and development: Morning Blossom Biotechnology Co., Ltd., Taipei, Taiwan), corn starch, crystalline cellulose and excipients in plant capsules.
  Interventions: Dietary Supplement: ExoBDNF SWP-CGPA01 (Pediococcus acidilactici)Capsules

INTERVENTIONS:
Dietary Supplement: ExoBDNF SWP-CGPA01 (Pediococcus acidilactici)Capsules — Product ingredients: microcrystalline cellulose, corn starch, SWP-CGPA01 Pediococcus acidilactici powder (1.0 x 10^10 CFU); Capsule shell composition: HPMC (hydroxypropyl methylcellulose), pure water, titanium dioxide, gelatin.

SUMMARY:
This open-label, single-group, pre/post-test clinical study was conducted to investigate whether ExoBDNF probiotic supplementation could improve cognitive ability. It is expected that 40 subjects aged 18 years and above will be recruited, with a target of 30 cases, to take ExoBDNF probiotics for a total of 8 weeks.

DETAILED DESCRIPTION:
Pre-test and post-test were conducted at week 0 and week 9, respectively. The test items included Cognitive Test Battery, SCD-Q Subjective Cognitive Decline Questionnaire, TCQ Cognitive Function Scale, MMSE Mini-Mental Scale, MoCA Montreal Cognitive Assessment Scale, PSQI Pittsburgh Sleep Quality Scale and DASS-21 Depression, Anxiety and Stress Scale, as well as blood biochemical examination and fecal intestinal flora analysis. The subjects were asked to take a capsule containing 1 x 1010 CFU of ExoBDNF probiotics once daily.

Subjects are required to maintain a regular lifestyle. After starting the diet, subjects filled out a daily diary that included questions about study product intake, other food intake, bowel movement frequency, stool quality (consistency and color), any medications received, and any unpleasant symptoms such as diarrhea, constipation, vomiting, flatulence, and discomfort. It is expected that this project will help clarify whether supplementation with Pediococcus acidilactici ExoBDNF can help improve cognitive ability, sleep or mental health.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be volunteers who are 18 years of age or older, mentally clear and able to communicate.
2. Subjects who agree to participate in this trial and voluntarily sign the trial consent form.

Exclusion Criteria:

1. Subjects who are expected to be or have been confirmed to be pregnant (medical history).
2. Subjects with gallbladder disease, gastrointestinal disease, gout, porphyria, or a history of gastric weight control surgery.
3. Subjects with high blood pressure (≥160/100 mmHg after resting for 10 minutes) or taking diuretics.
4. Subjects with heart disease, hepatorenal insufficiency, hyperthyroidism or hypothyroidism, Cushing's syndrome, malignant tumors, or any other disease that may affect the results of the study.
5. Subjects with severe hearing or visual impairment that makes it impossible to perform examinations and assessments.
6. Subjects with any history of brain surgery, penetrating, neurovascular, infectious or other severe brain injury, epilepsy or other major neurological abnormalities, such as traumatic brain injury with loss of consciousness for more than 24 hours, or memory loss after head trauma for more than 7 days were excluded.
7. Subjects with intellectual disabilities.
8. Subjects who had consumed probiotics or were expected to consume probiotics within 2 weeks before the screening visit.
9. Subjects who had participated in or were expected to participate in clinical trials within 4 weeks before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Cognitive Decline Questionnaire (SCD-Q) scale | 8 weeks
  To compare whether there is a statistically significant difference in the Subjective Cognitive Decline Questionnaire (SCD-Q) scale scores between the trial group and the placebo group after taking the probiotics for 8 weeks compared with the values 8 weeks ago (baseline).

SECONDARY OUTCOMES:
Computerized cognitive test-Go/No go | 8 weeks
  Mainly used to assess concentration, reaction and memory, this task is used to measure the brain's ability to distinguish relevant and irrelevant information. The task requires participants to pay attention to the prompt and judge whether the subsequent stimulus is the target.
Computerized cognitive test-Task-switching | 8 weeks
  Mainly used to assess the brain's task switching ability, the task switching task is used to measure the flexibility of selective attention. The task requires participants to switch their attention between judging the cardinality of even numbers or the size of numbers.
Computerized cognitive test-Working memory | 8 weeks
  Mainly used to assess memory, this working memory task refers to the spatial span task (Corsi block tapping task), which is used to measure spatial short-term memory capacity.
Depression Anxiety Stress Scale DASS-21 | 8 weeks
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-assessment questionnaire that assesses sleep quality and sleep disturbances over a one-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, MD, Principal Investigator — Director, Child and Adolescent Psychiatry, Department of Psychiatry
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lequesne M, Cassan P, Nallet J, Ryckewaert A, de Seze S. [Vertebral hyperostosis and diabetes mellitus]. Rev Rhum Mal Osteoartic. 1970 Apr;37(4):281-6. No abstract available. French. PMID 5448694
- [Result] Erickson KI, Donofry SD, Sewell KR, Brown BM, Stillman CM. Cognitive Aging and the Promise of Physical Activity. Annu Rev Clin Psychol. 2022 May 9;18:417-442. doi: 10.1146/annurev-clinpsy-072720-014213. Epub 2022 Jan 19. PMID 35044793
- [Result] O'Donoghue MC, Murphy SE, Zamboni G, Nobre AC, Mackay CE. APOE genotype and cognition in healthy individuals at risk of Alzheimer's disease: A review. Cortex. 2018 Jul;104:103-123. doi: 10.1016/j.cortex.2018.03.025. Epub 2018 Mar 30. PMID 29800787
- [Result] Shakersain B, Santoni G, Larsson SC, Faxen-Irving G, Fastbom J, Fratiglioni L, Xu W. Prudent diet may attenuate the adverse effects of Western diet on cognitive decline. Alzheimers Dement. 2016 Feb;12(2):100-109. doi: 10.1016/j.jalz.2015.08.002. Epub 2015 Sep 3. PMID 26342761
- [Result] Schneider S, Wright CM, Heuckeroth RO. Unexpected Roles for the Second Brain: Enteric Nervous System as Master Regulator of Bowel Function. Annu Rev Physiol. 2019 Feb 10;81:235-259. doi: 10.1146/annurev-physiol-021317-121515. Epub 2018 Oct 31. PMID 30379617
- [Result] Kowalski K, Mulak A. Brain-Gut-Microbiota Axis in Alzheimer's Disease. J Neurogastroenterol Motil. 2019 Jan 31;25(1):48-60. doi: 10.5056/jnm18087. PMID 30646475
- [Result] D'Amato A, Di Cesare Mannelli L, Lucarini E, Man AL, Le Gall G, Branca JJV, Ghelardini C, Amedei A, Bertelli E, Regoli M, Pacini A, Luciani G, Gallina P, Altera A, Narbad A, Gulisano M, Hoyles L, Vauzour D, Nicoletti C. Faecal microbiota transplant from aged donor mice affects spatial learning and memory via modulating hippocampal synaptic plasticity- and neurotransmission-related proteins in young recipients. Microbiome. 2020 Oct 1;8(1):140. doi: 10.1186/s40168-020-00914-w. PMID 33004079
- [Result] Dominguez LJ, Barbagallo M. Nutritional prevention of cognitive decline and dementia. Acta Biomed. 2018 Jun 7;89(2):276-290. doi: 10.23750/abm.v89i2.7401. PMID 29957766
- [Result] Forsythe P, Bienenstock J, Kunze WA. Vagal pathways for microbiome-brain-gut axis communication. Adv Exp Med Biol. 2014;817:115-33. doi: 10.1007/978-1-4939-0897-4_5. PMID 24997031
- [Result] Sampson TR, Mazmanian SK. Control of brain development, function, and behavior by the microbiome. Cell Host Microbe. 2015 May 13;17(5):565-76. doi: 10.1016/j.chom.2015.04.011. PMID 25974299
- [Result] Sharon G, Garg N, Debelius J, Knight R, Dorrestein PC, Mazmanian SK. Specialized metabolites from the microbiome in health and disease. Cell Metab. 2014 Nov 4;20(5):719-730. doi: 10.1016/j.cmet.2014.10.016. Epub 2014 Nov 4. PMID 25440054
- [Result] Liu N, Yang D, Sun J, Li Y. Probiotic supplements are effective in people with cognitive impairment: a meta-analysis of randomized controlled trials. Nutr Rev. 2023 Aug 10;81(9):1091-1104. doi: 10.1093/nutrit/nuac113. PMID 36629438
- [Result] Fei Y, Wang R, Lu J, Peng S, Yang S, Wang Y, Zheng K, Li R, Lin L, Li M. Probiotic intervention benefits multiple neural behaviors in older adults with mild cognitive impairment. Geriatr Nurs. 2023 May-Jun;51:167-175. doi: 10.1016/j.gerinurse.2023.03.006. Epub 2023 Mar 28. PMID 36990042
- [Result] Chong HX, Yusoff NAA, Hor YY, Lew LC, Jaafar MH, Choi SB, Yusoff MSB, Wahid N, Abdullah MFIL, Zakaria N, Ong KL, Park YH, Liong MT. Lactobacillus plantarum DR7 alleviates stress and anxiety in adults: a randomised, double-blind, placebo-controlled study. Benef Microbes. 2019 Apr 19;10(4):355-373. doi: 10.3920/BM2018.0135. Epub 2019 Mar 18. PMID 30882244
- [Result] Kobayashi Y, Kinoshita T, Matsumoto A, Yoshino K, Saito I, Xiao JZ. Bifidobacterium Breve A1 Supplementation Improved Cognitive Decline in Older Adults with Mild Cognitive Impairment: An Open-Label, Single-Arm Study. J Prev Alzheimers Dis. 2019;6(1):70-75. doi: 10.14283/jpad.2018.32. PMID 30569089
- [Result] Adolphe M, Sawayama M, Maurel D, Delmas A, Oudeyer PY, Sauzeon H. An Open-Source Cognitive Test Battery to Assess Human Attention and Memory. Front Psychol. 2022 Jun 10;13:880375. doi: 10.3389/fpsyg.2022.880375. eCollection 2022. PMID 35756204
- [Result] Yen YC, Chiu NY, Hwang TJ, Su TP, Yang YK, Chen CS, Li CT, Su KP, Lai TJ, Chang CM. A Multi-Center Study for the Development of the Taiwan Cognition Questionnaire (TCQ) in Major Depressive Disorder. J Pers Med. 2022 Feb 26;12(3):359. doi: 10.3390/jpm12030359. PMID 35330360
- [Result] Tsai CL, Chou KH, Lee PL, Liang CS, Kuo CY, Lin GY, Lin YK, Hsu YC, Ko CA, Yang FC, Lin CP. Shared alterations in hippocampal structural covariance in subjective cognitive decline and migraine. Front Aging Neurosci. 2023 Jun 20;15:1191991. doi: 10.3389/fnagi.2023.1191991. eCollection 2023. PMID 37409010
- [Result] de Oliveira BH, Lins EF, Kunde NF, Salgado ASI, Martins LM, Bobinski F, Vieira WF, Cassano P, Quialheiro A, Martins DF. Transcranial photobiomodulation increases cognition and serum BDNF levels in adults over 50 years: A randomized, double-blind, placebo-controlled trial. J Photochem Photobiol B. 2024 Nov;260:113041. doi: 10.1016/j.jphotobiol.2024.113041. Epub 2024 Oct 5. PMID 39423445
- [Result] Nilsson P, Saito T, Saido TC. New mouse model of Alzheimer's. ACS Chem Neurosci. 2014 Jul 16;5(7):499-502. doi: 10.1021/cn500105p. Epub 2014 May 22. PMID 24852598
- [Result] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123